CLINICAL TRIAL: NCT02135341
Title: Comparative Study of Safety and Efficacy Between 100 U Suburothelial Injection and 50 U Suburothelial Plus 50 U Urethral Injections of Botulinum Toxin A in Treatment of Patients With Detrusor Overactivity and Impaired Contractility
Brief Title: Injections of Botulinum Toxin A in Treatment of Patients With Detrusor Overactivity and Impaired Contractility
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Buddhist Tzu Chi General Hospital (Other)
Responsible Party: Principal Investigator, Hann-Chorng Kuo, Director of Urology, Buddhist Tzu Chi General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TCGHUROL010
Record Dates: First submitted 2014-05-08; First posted 2014-05-09 (Estimated); Last update posted 2017-02-15 (Actual); Status verified 2017-02

CONDITIONS: Botulinum Toxins, Type A
Keywords: Detrusor Overactivity; Impaired Contractility; Botulinum Toxin A (BoNT-A)
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Botulinum Toxins, Type A; incobotulinumtoxinA

STUDY DESIGN:
Intervention Model Description: Patients with urodynamically proven DHIC and age-matched controlled OAB patients with urodynamic DO selected from our previous clinical trials were compared for the treatment outcome of onabotulinumtoxinA injection
Masking Description: No masking was designed in this study
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A: Botulinum toxin A (Experimental): BoNT-A 100 units in normal saline 10ml, suburothelial injection at 20 sites of bladder wall in single treatment
  Interventions: Drug: Botulinum toxin A
- Group B: Botulinum toxin A (Experimental): BoNT-A 100 units in normal saline 10ml, suburothelial injection 50 U in 10 sites and 50 U urethral injections in 5 sites
  Interventions: Drug: Botulinum toxin A

INTERVENTIONS:
Drug: Botulinum toxin A — BoNT-A 100 units in normal saline 10ml, suburothelial injection at 20 sites of bladder wall in single treatment
  Other Names: BoNT-A; BOTOX (Allergan, Irvine, CA, USA)
  Arms: Group A: Botulinum toxin A
Drug: Botulinum toxin A — BoNT-A 100 units in normal saline 10ml, suburothelial injection 50 U in 10 sites and 50 U urethral injections in 5 sites
  Other Names: BoNT-A; BOTOX (Allergan, Irvine, CA, USA)
  Arms: Group B: Botulinum toxin A

SUMMARY:
The objectives of this study is to evaluate and compare the efficacy and safety between 100 U of botulinum toxin A (BoNT-A) suburothelial injections and combined 50 U of BoNT-A suburothelial injections and 50 U urethral injection for the treatment of detrusor overactivity and inadequate contractility (DHIC) refractory to antimuscarinic agents

DETAILED DESCRIPTION:
Overactive bladder (OAB) is a symptom syndrome characterized by urgency frequency with or without urgency incontinence, usually no metabolic or anatomical disorders can be found and it may have great impact on quality of life. OAB symptoms were found to have a significant effect on the emotional well-being and productivity of those affected. Although there are several new therapeutic options with promising treatment outcome, antimuscarinic drugs remain the first line treatment and clinical effects with good tolerability have been confirmed. However, not all OAB patients can benefit from antimuscarinic agent, and this treatment has some adverse effects such as dizziness, dry mouth, blurred vision, and constipation, which are intolerable for some patients. Of these patients intravesical botulinum toxin (BoNT) injections provide an alternative treatment with a favorable efficacy.

Based on the understanding of the pathophysiology of OAB and detrusor overactivity (DO), BoNT has been enthusiastically applied in treating urinary urgency or incontinence refractory to antimuscarinics in recent years. Although promising therapeutic effects have been confirmed by several case series or clinical trials, the occurrence of adverse events are reported inconsistently. Analysis of patients demographics and urodynamic variables reveals that patients with ageing, low detrusor contractility, with chronic medical disease carry risks of adverse events. Although safety and efficacy were similar between elderly patients without frailty and younger patients, an increased risk of large post-void residual urine volume and a lower long-term success rate in frail elderly patients were noted after intravesical 100 U BoNT-A injection for refractory idiopathic DO. Therefore, careful dose and injection site adjustment and patient selection is mandatory to achieve satisfactory results using intravesical BoNT-A therapy.

This study aimed at compare the safety and efficacy between 100 U suburothelial injection and combined 50 U suburothelial and 50 U urethral sphincter injection of BoNT-A in patients with detrusor overactivity and inadequate contractility (DHIC). A total of 60 patients with DHIC will be enrolled and randomly allocated to each group and treated with either regimen. The safety and efficacy will be assessed by the Patient's Perception of Bladder Condition (PPBC) at different time points after injection. The results of this study may provide valuable evidence for the rational treatment regimen for patients with DHIC.

Estimated Total Sample Size 60 evaluable patients in total will be recruited

Method of Patient Assignment

Patients who meet all eligible requirements for entry into the study will be randomized into one of the two treatment groups in 1:1 ratio as shown below:

1. BoNT-A 100 units in normal saline 10ml, suburothelial injection at 20 sites of bladder wall in single treatment
2. BoNT-A 100 units in normal saline 10ml, suburothelial injection 50 U in 10 sites and 50 U urethral injections in 5 sites

Patient Inclusion Criteria

1. Adults with age of 20 years old or above
2. Patients with symptoms of urgency frequency and/or urge incontinence and urodynamically proven DHIC (defined by the International Continence Society (ICS) recommendation as: spontaneous detrusor contraction occurring during bladder filling phase or occurring before uninhibited detrusor contraction voiding at bladder capacity of less than 350ml in the urodynamic study, and has postvoid residual of more than 100ml but less than 250ml)
3. Free of active urinary tract infection
4. Free of bladder outlet obstruction on enrollment
5. Free of overt neurogenic bladder dysfunction
6. Having been treated with antimuscarinic agents for at least 1 months without effect or with intolerable adverse effects
7. Patient or his/her legally acceptable representative has signed the written informed consent form

Patient Exclusion Criteria

1. Use of antimuscarinic agent and effective in treatment of lower urinary tract symptoms
2. Patients with severe cardiopulmonary disease and such as congestive heart failure, arrhythmia, poorly controlled hypertension, not able to receive regular follow-up
3. Patients with bladder outlet obstruction on enrollment
4. Patients with postvoid residual > 250ml
5. Patients with uncontrolled confirmed diagnosis of acute urinary tract infection
6. Patients have laboratory abnormalities at screening including:

   Alanine aminotransferase (ALT)> 3 x upper limit of normal range Aspartate aminotransferase (AST)> 3 x upper limit of normal range Patients have abnormal serum creatinine level > 2 x upper limit of normal range
7. Patients with any contraindication to be urethral catheterization during treatment
8. Patients with any other serious disease considered by the investigator not in the condition to enter the trial
9. Patients participated investigational drug trial within 1 month before entering this study

Data Analysis The efficacy evaluation will be performed on intention-to-treat populations (ITT) and per-protocol populations (PPP) datasets while the safety evaluation will be performed on ITT datasets. The primary conclusion will be made for the primary endpoint and secondary endpoint on the ITT population..

Efficacy Endpoint Analysis Net change of each efficacy item will be analyzed by paired t-test between baseline and post-treatment in the treatment group and controlled group. The net changes of each efficacy item will be analyzed by ANOVA test to compare between treatment group and controlled group. The global assessment by the patients will be analyzed by chi-square test between the treatment and controlled group.

All efficacy variables will be reported of respective point estimated and 95% confidence interval. Comparison tests will be reported of respective p value.

Safety Endpoints Adverse events will be reported by both controlled and treatment groups and by physiological systems as appropriate. Incidence of adverse events and the categories of adverse event severity between treatments will be analyzed by Cochran-Mantel-Haenszel test. The coding system used will be the Coding Symbols for a Thesaurus of Adverse Reaction Terms (COSTART).

Changes in physical examinations will be displayed for each individual system. All statistical tests used will be two-tailed with α= 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Adults with age of 20 years old or above
* Patients with symptoms of urgency frequency and/or urge incontinence and urodynamically proven DHIC (defined by the ICS recommendation as: spontaneous detrusor contraction occurring during bladder filling phase or occurring before uninhibited detrusor contraction voiding at bladder capacity of less than 350ml in the urodynamic study, and has postvoid residual of more than 100ml but less than 250ml)
* Free of active urinary tract infection
* Free of bladder outlet obstruction on enrollment
* Free of overt neurogenic bladder dysfunction
* Having been treated with antimuscarinic agents for at least 1 months without effect or with intolerable adverse effects
* Patient or his/her legally acceptable representative has signed the written informed consent form

Exclusion Criteria:

* Use of antimuscarinic agent and effective in treatment of lower urinary tract symptoms
* Patients with severe cardiopulmonary disease and such as congestive heart failure, arrhythmia, poorly controlled hypertension, not able to receive regular follow-up
* Patients with bladder outlet obstruction on enrollment
* Patients with postvoid residual > 250ml
* Patients with uncontrolled confirmed diagnosis of acute urinary tract infection
* Patients have laboratory abnormalities at screening including:

ALT> 3 x upper limit of normal range AST> 3 x upper limit of normal range Patients have abnormal serum creatinine level > 2 x upper limit of normal range

* Patients with any contraindication to be urethral catheterization during treatment
* Patients with any other serious disease considered by the investigator not in the condition to enter the trial
* Patients participated investigational drug trial within 1 month before entering this study

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Net change of the Patients Perception of Bladder Condition (PPBC) | Baseline and 3 months
  Net change of the Patients Perception of Bladder Condition (PPBC, scored from 1 to 6) from baseline to 3 months after the treatment day.
  Safety:
  1. Local adverse event incidences (hematuria, micturition pain, urinary tract infection (UTI), urinary retention)
  2. Systemic adverse events.
  Safety:
  Systemic adverse events

SECONDARY OUTCOMES:
Net change of the International Prostate Symptom Score (IPSS) | Baseline and 3 months
  Net change of the following parameters from baseline to 3 month after the treatment day: lower urinary tract symptom score (including empty and storage IPSS)
Net change of the bladder capacity | Baseline and 3 months
  Efficacy:
  Net change of the following parameters from baseline to 3 month after the treatment day: bladder capacity
  Safety:
  Local adverse event incidences (hematuria, micturition pain, UTI, urinary retention) Systemic adverse events.
Net change of the voiding frequency at daytime | Baseline and 3 months
  Efficacy:
  Net change of the following parameters from baseline to 3 month after the treatment day: voiding frequency at daytime.
  Safety:
  Local adverse event incidences (hematuria, micturition pain, UTI, urinary retention) Systemic adverse events.
Net change of the voiding frequency at night time | Baseline and 3 months
  Efficacy:
  Net change of the following parameters from baseline to 3 month after the treatment day: voiding frequency at night time.
  Safety:
  Local adverse event incidences (hematuria, micturition pain, UTI, urinary retention) Systemic adverse events.
Net change of voiding urgency severity score | Baseline and 3 months
  Efficacy:
  Net change of the following parameters from baseline to 3 month after the treatment day: urgency severity score
  Safety:
  Local adverse event incidences (hematuria, micturition pain, UTI, urinary retention) Systemic adverse events.
Net change of the first sensation of bladder filling | Baseline and 3 months
  Efficacy:
  Net change of the urodynamic parameters: first sensation of bladder filling from baseline to 3 months after the treatment day.
  Safety:
  Local adverse event incidences (hematuria, micturition pain, UTI, urinary retention) Systemic adverse events.
Net change of the urge sensation | Baseline and 3 months
  Efficacy:
  Net change of the urodynamic parameters: urge sensation from baseline to 3 months after the treatment day.
  Safety:
  Local adverse event incidences (hematuria, micturition pain, UTI, urinary retention) Systemic adverse events.
Net change of the presence of detrusor overactivity | Baseline and 3 months
  Efficacy:
  Net change of the urodynamic parameters: presence of detrusor overactivity from baseline to 3 months after the treatment day.
  Safety:
  Local adverse event incidences (hematuria, micturition pain, UTI, urinary retention) Systemic adverse events.
Net change of the cystometric bladder capacity | Baseline and 3 months
  Efficacy:
  Net change of the urodynamic parameters: cystometric bladder capacity from baseline to 3 months after the treatment day.
  Safety:
  Local adverse event incidences (hematuria, micturition pain, UTI, urinary retention) Systemic adverse events.
Net change of the first sensation of detrusor pressure | Baseline and 3 months
  Efficacy:
  Net change of the urodynamic parameters: detrusor pressure from baseline to 3 months after the treatment day.
  Safety:
  Local adverse event incidences (hematuria, micturition pain, UTI, urinary retention) Systemic adverse events.
Net change of the first sensation of bladder compliance | Baseline and 3 months
  Efficacy:
  Net change of the urodynamic parameters: bladder compliance from baseline to 3 months after the treatment day.
  Safety:
  Local adverse event incidences (hematuria, micturition pain, UTI, urinary retention) Systemic adverse events.
Net change of the maximum flow rate | Baseline and 3 months
  Efficacy:
  Net change of the urodynamic parameters: maximum flow rate from baseline to 3 months after the treatment day.
  Safety:
  Local adverse event incidences (hematuria, micturition pain, UTI, urinary retention) Systemic adverse events.
Net change of the first sensation of voided volume | Baseline and 3 months
  Efficacy:
  Net change of the urodynamic parameters: voided volume from baseline to 3 months after the treatment day.
  Safety:
  Local adverse event incidences (hematuria, micturition pain, UTI, urinary retention) Systemic adverse events.
Net change of the postvoid residual volume | Baseline and 3 months
  Efficacy:
  Net change of the urodynamic parameters: postvoid residual volume from baseline to 3 months after the treatment day.
  Safety:
  Local adverse event incidences (hematuria, micturition pain, UTI, urinary retention) Systemic adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Hann-Chorng Kuo, M.D., Principal Investigator — Department of Urology, Buddhist Tzu Chi General Hospital and Tzu Chi University
Locations (1):
- Buddhist Tzu Chi General Hospital, Hualien City, Taiwan

IPD SHARING:
Plan to Share IPD: No
No IPD is planned to share

REFERENCES:
- [Background] Abrams P, Kelleher CJ, Kerr LA, Rogers RG. Overactive bladder significantly affects quality of life. Am J Manag Care. 2000 Jul;6(11 Suppl):S580-90. PMID 11183901
- [Background] Irwin DE, Milsom I, Kopp Z, Abrams P, Cardozo L. Impact of overactive bladder symptoms on employment, social interactions and emotional well-being in six European countries. BJU Int. 2006 Jan;97(1):96-100. doi: 10.1111/j.1464-410X.2005.05889.x. PMID 16336336
- [Background] Yoshimura N. Lower urinary tract symptoms (LUTS) and bladder afferent activity. Neurourol Urodyn. 2007 Oct;26(6 Suppl):908-13. doi: 10.1002/nau.20487. PMID 17654565
- [Background] Chapple CR. Muscarinic receptor antagonists in the treatment of overactive bladder. Urology. 2000 May;55(5A Suppl):33-46; discussion 50. doi: 10.1016/s0090-4295(99)00492-6. PMID 10767450
- [Background] Kuo HC. Urodynamic evidence of effectiveness of botulinum A toxin injection in treatment of detrusor overactivity refractory to anticholinergic agents. Urology. 2004 May;63(5):868-72. doi: 10.1016/j.urology.2003.12.007. PMID 15134967
- [Background] Kessler TM, Danuser H, Schumacher M, Studer UE, Burkhard FC. Botulinum A toxin injections into the detrusor: an effective treatment in idiopathic and neurogenic detrusor overactivity? Neurourol Urodyn. 2005;24(3):231-6. doi: 10.1002/nau.20105. PMID 15747344
- [Background] Werner M, Schmid DM, Schussler B. Efficacy of botulinum-A toxin in the treatment of detrusor overactivity incontinence: a prospective nonrandomized study. Am J Obstet Gynecol. 2005 May;192(5):1735-40. doi: 10.1016/j.ajog.2004.11.052. PMID 15902187
- [Background] Kuo HC. Clinical effects of suburothelial injection of botulinum A toxin on patients with nonneurogenic detrusor overactivity refractory to anticholinergics. Urology. 2005 Jul;66(1):94-8. doi: 10.1016/j.urology.2005.02.002. PMID 15992869
- [Background] Schulte-Baukloh H, Weiss C, Stolze T, Sturzebecher B, Knispel HH. Botulinum-A toxin for treatment of overactive bladder without detrusor overactivity: urodynamic outcome and patient satisfaction. Urology. 2005 Jul;66(1):82-7. doi: 10.1016/j.urology.2005.01.036. PMID 15992872
- [Background] Schulte-Baukloh H, Weiss C, Stolze T, Herholz J, Sturzebecher B, Miller K, Knispel HH. Botulinum-A toxin detrusor and sphincter injection in treatment of overactive bladder syndrome: objective outcome and patient satisfaction. Eur Urol. 2005 Dec;48(6):984-90; discussion 990. doi: 10.1016/j.eururo.2005.06.021. Epub 2005 Jul 18. PMID 16126328
- [Background] Ghei M, Maraj BH, Miller R, Nathan S, O'Sullivan C, Fowler CJ, Shah PJ, Malone-Lee J. Effects of botulinum toxin B on refractory detrusor overactivity: a randomized, double-blind, placebo controlled, crossover trial. J Urol. 2005 Nov;174(5):1873-7; discussion 1877. doi: 10.1097/01.ju.0000177477.83991.88. PMID 16217327
- [Background] Rajkumar GN, Small DR, Mustafa AW, Conn G. A prospective study to evaluate the safety, tolerability, efficacy and durability of response of intravesical injection of botulinum toxin type A into detrusor muscle in patients with refractory idiopathic detrusor overactivity. BJU Int. 2005 Oct;96(6):848-52. doi: 10.1111/j.1464-410X.2005.05725.x. PMID 16153215
- [Background] Popat R, Apostolidis A, Kalsi V, Gonzales G, Fowler CJ, Dasgupta P. A comparison between the response of patients with idiopathic detrusor overactivity and neurogenic detrusor overactivity to the first intradetrusor injection of botulinum-A toxin. J Urol. 2005 Sep;174(3):984-9. doi: 10.1097/01.ju.0000169480.43557.31. PMID 16094019
- [Background] Kuo HC. Will suburothelial injection of small dose of botulinum A toxin have similar therapeutic effects and less adverse events for refractory detrusor overactivity? Urology. 2006 Nov;68(5):993-7; discussion 997-8. doi: 10.1016/j.urology.2006.05.054. PMID 17113890
- [Background] Schmid DM, Sauermann P, Werner M, Schuessler B, Blick N, Muentener M, Strebel RT, Perucchini D, Scheiner D, Schaer G, John H, Reitz A, Hauri D, Schurch B. Experience with 100 cases treated with botulinum-A toxin injections in the detrusor muscle for idiopathic overactive bladder syndrome refractory to anticholinergics. J Urol. 2006 Jul;176(1):177-85. doi: 10.1016/S0022-5347(06)00590-8. PMID 16753396
- [Background] Lucioni A, Rapp DE, Gong EM, Fedunok P, Bales GT. Intravesical botulinum type A toxin injection in patients with overactive bladder: Trigone versus trigone-sparing injection. Can J Urol. 2006 Oct;13(5):3291-5. PMID 17076955
- [Background] Hoebeke P, De Caestecker K, Vande Walle J, Dehoorne J, Raes A, Verleyen P, Van Laecke E. The effect of botulinum-A toxin in incontinent children with therapy resistant overactive detrusor. J Urol. 2006 Jul;176(1):328-30; discussion 330-1. doi: 10.1016/S0022-5347(06)00301-6. PMID 16753434
- [Background] Kalsi V, Apostolidis A, Popat R, Gonzales G, Fowler CJ, Dasgupta P. Quality of life changes in patients with neurogenic versus idiopathic detrusor overactivity after intradetrusor injections of botulinum neurotoxin type A and correlations with lower urinary tract symptoms and urodynamic changes. Eur Urol. 2006 Mar;49(3):528-35. doi: 10.1016/j.eururo.2005.12.012. Epub 2006 Jan 6. PMID 16426735
- [Background] Hirst GR, Watkins AJ, Guerrero K, Wareham K, Emery SJ, Jones DR, Lucas MG. Botulinum toxin B is not an effective treatment of refractory overactive bladder. Urology. 2007 Jan;69(1):69-73. doi: 10.1016/j.urology.2006.09.005. PMID 17270619
- [Background] Ghalayini IF, Al-Ghazo MA. Intradetrusor injection of botulinum-A toxin in patients with idiopathic and neurogenic detrusor overactivity: urodynamic outcome and patient satisfaction. Neurourol Urodyn. 2007;26(4):531-536. doi: 10.1002/nau.20403. PMID 17330289
- [Background] Sahai A, Khan MS, Dasgupta P. Efficacy of botulinum toxin-A for treating idiopathic detrusor overactivity: results from a single center, randomized, double-blind, placebo controlled trial. J Urol. 2007 Jun;177(6):2231-6. doi: 10.1016/j.juro.2007.01.130. PMID 17509328
- [Background] Kuo HC. Comparison of effectiveness of detrusor, suburothelial and bladder base injections of botulinum toxin a for idiopathic detrusor overactivity. J Urol. 2007 Oct;178(4 Pt 1):1359-63. doi: 10.1016/j.juro.2007.05.136. Epub 2007 Aug 16. PMID 17706718
- [Background] Jeffery S, Fynes M, Lee F, Wang K, Williams L, Morley R. Efficacy and complications of intradetrusor injection with botulinum toxin A in patients with refractory idiopathic detrusor overactivity. BJU Int. 2007 Dec;100(6):1302-6. doi: 10.1111/j.1464-410X.2007.07186.x. PMID 17979928
- [Background] Karsenty G, Elzayat E, Delapparent T, St-Denis B, Lemieux MC, Corcos J. Botulinum toxin type a injections into the trigone to treat idiopathic overactive bladder do not induce vesicoureteral reflux. J Urol. 2007 Mar;177(3):1011-4. doi: 10.1016/j.juro.2006.10.047. PMID 17296399
- [Background] Kalsi V, Apostolidis A, Gonzales G, Elneil S, Dasgupta P, Fowler CJ. Early effect on the overactive bladder symptoms following botulinum neurotoxin type A injections for detrusor overactivity. Eur Urol. 2008 Jul;54(1):181-7. doi: 10.1016/j.eururo.2007.12.029. Epub 2007 Dec 26. PMID 18191323
- [Background] Kuschel S, Werner M, Schmid DM, Faust E, Schuessler B. Botulinum toxin-A for idiopathic overactivity of the vesical detrusor: a 2-year follow-up. Int Urogynecol J Pelvic Floor Dysfunct. 2008 Jul;19(7):905-9. doi: 10.1007/s00192-007-0548-9. Epub 2008 Jan 19. PMID 18204796
- [Background] Brubaker L, Richter HE, Visco A, Mahajan S, Nygaard I, Braun TM, Barber MD, Menefee S, Schaffer J, Weber AM, Wei J; Pelvic Floor Disorders Network. Refractory idiopathic urge urinary incontinence and botulinum A injection. J Urol. 2008 Jul;180(1):217-22. doi: 10.1016/j.juro.2008.03.028. Epub 2008 May 21. PMID 18499184
- [Background] White WM, Pickens RB, Doggweiler R, Klein FA. Short-term efficacy of botulinum toxin a for refractory overactive bladder in the elderly population. J Urol. 2008 Dec;180(6):2522-6. doi: 10.1016/j.juro.2008.08.030. Epub 2008 Oct 19. PMID 18930481
- [Background] Khan S, Kessler TM, Apostolidis A, Kalsi V, Panicker J, Roosen A, Gonzales G, Haslam C, Elneil S, Fowler CJ, Dasgupta P. What a patient with refractory idiopathic detrusor overactivity should know about botulinum neurotoxin type a injection. J Urol. 2009 Apr;181(4):1773-8. doi: 10.1016/j.juro.2008.11.110. Epub 2009 Feb 23. PMID 19233414
- [Background] Cohen BL, Barboglio P, Rodriguez D, Gousse AE. Preliminary results of a dose-finding study for botulinum toxin-A in patients with idiopathic overactive bladder: 100 versus 150 units. Neurourol Urodyn. 2009;28(3):205-8. doi: 10.1002/nau.20611. PMID 19058190
- [Background] Sahai A, Sangster P, Kalsi V, Khan MS, Fowler CJ, Dasgupta P. Assessment of urodynamic and detrusor contractility variables in patients with overactive bladder syndrome treated with botulinum toxin-A: is incomplete bladder emptying predictable? BJU Int. 2009 Mar;103(5):630-4. doi: 10.1111/j.1464-410X.2008.08076.x. Epub 2008 Oct 16. PMID 18990156
- [Background] Flynn MK, Amundsen CL, Perevich M, Liu F, Webster GD. Outcome of a randomized, double-blind, placebo controlled trial of botulinum A toxin for refractory overactive bladder. J Urol. 2009 Jun;181(6):2608-15. doi: 10.1016/j.juro.2009.01.117. Epub 2009 Apr 16. PMID 19375091
- [Background] Kessler TM, Khan S, Panicker J, Roosen A, Elneil S, Fowler CJ. Clean intermittent self-catheterization after botulinum neurotoxin type A injections: short-term effect on quality of life. Obstet Gynecol. 2009 May;113(5):1046-1051. doi: 10.1097/AOG.0b013e3181a1f5ea. PMID 19384119
- [Background] Kuo HC, Liao CH, Chung SD. Adverse events of intravesical botulinum toxin a injections for idiopathic detrusor overactivity: risk factors and influence on treatment outcome. Eur Urol. 2010 Dec;58(6):919-26. doi: 10.1016/j.eururo.2010.09.007. Epub 2010 Sep 17. PMID 20864251
- [Background] Liao CH, Kuo HC. Increased risk of large post-void residual urine and decreased long-term success rate after intravesical onabotulinumtoxinA injection for refractory idiopathic detrusor overactivity. J Urol. 2013 May;189(5):1804-10. doi: 10.1016/j.juro.2012.11.089. Epub 2012 Nov 20. PMID 23178902